CLINICAL TRIAL: NCT06084715
Title: Impact of Nutritional Support for Tuberculosis on Intermediate and Terminal Undernutrition and Treatment Outcomes: the INSTITUT Study
Brief Title: The INSTITUT Study Tuberculosis Nutritional Support
Acronym: INSTITUT
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: The International Union Against Tuberculosis and Lung Disease (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-43096
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pulmonary; Undernutrition
Keywords: Persons with TB (PWTB); Nutritional support; Republic of Benin; Togolese Republic; Treatment failure; TB relapse; Chronic obstructive pulmonary disease (COPD); Quality of life
MeSH Terms: conditions — Tuberculosis, Pulmonary; Malnutrition; Pulmonary Disease, Chronic Obstructive | interventions — Nutritional Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nutritional support group: Participants in this group will be enrolled in Benin and will receive nutritional support from the hospital where they receive care. They will be followed for 12 months.
  Interventions: Other: Nutritional support
- Standard of care group: Participants in this group will be enrolled in Togo and will not receive nutritional support from the hospital where they receive care. They will be followed for 12 months.

INTERVENTIONS:
Other: Nutritional support — The hospitals in Benin already provide nutritional support for patients with pulmonary TB which will continue throughout the study.
  Groups: Nutritional support group

SUMMARY:
Undernutrition is a leading global risk factor of tuberculosis (TB) and a prevalent comorbidity associated with TB. In Benin, the National TB Program systematically provides nutritional support to all persons with TB (PWTB), distributing prepared foods to hospitalized patients and food baskets during outpatient care. In Togo, the PWTB population is similar to that of Benin; however, Togo does not have a systematic program in place to provide nutritional support to these patients.

The investigators will perform a prospective cohort analysis using anonymized TB patient data from the National TB Programs of Benin and Togo. Participants enrolled in Benin will receive nutritional support from the hospital while those enrolled in Togo will not. Participants in Togo who do not receive nutritional support will serve as a control. Unfavorable outcomes in both groups such as treatment failure, death, or relapse will be compared. The results from this study should help to shape TB programs in the future by incorporating nutritional support.

DETAILED DESCRIPTION:
The objectives of this prospective cohort analysis are:

* To estimate the impact of nutritional support on TB treatment outcomes
* To estimate the impact of nutritional support on the nutritional status of persons with TB (PWTB) at the end of treatment.

Pulmonary TB patients who meet eligibility criteria including being diagnosed with a smear-positive (>/=1+ AFB) and provide informed consent will be enrolled. A projected sample of 1050 participants will be enrolled and followed for approximately 12 months. 700 will be enrolled in Benin and 350 in Togo. Participants enrolled in Benin will receive nutritional support from the hospital while those enrolled in Togo will not.

Sputum samples will be collected at baseline and month two to confirm diagnosis and resolution of disease. Chest X-rays will be taken at enrollment, if not available by the TB program, and repeated 6 months following the end of TB treatment to assess for post-TB chronic lung disease. At all visits, surveys will be administered to assess for response to treatment and functional and economic recovery.

ELIGIBILITY:
Inclusion Criteria:

* Drug susceptible, Xpert [polymerase chain reaction (PCR) test for TB] positive and/or sputum stain positive for AFB (≥1+)
* Willing to attend follow-up visits and undergo study procedures

Exclusion Criteria:

* Drug resistant TB
* Has received 7 or more days of antimicrobial therapy
* Based on study staff observation, the participant is too sick to enroll. Defined as a score of 4 on the World Health Organization (WHO) Performance assessment.
* Pregnancy at the time of enrollment
* Individuals who are unable to participate in the 6-minute walk test due to pre-existing mobility issues due to disability, trauma, neurological compromise, or cardiopulmonary issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1050 participants will be enrolled and followed for approximately 12 months. 700 will be enrolled in Benin and 350 in Togo. Participants enrolled in Benin will receive nutritional support from the hospital while those enrolled in Togo will not.
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
Percent of participants with an unfavorable outcome | 12 months
  An unfavorable outcome will be a composite of TB treatment failure, death, or relapse based on patient evaluation 6 months after treatment completion.

SECONDARY OUTCOMES:
Number of participants with failure of sputum conversion | 2 months
  Failure for those with positive sputum smears at treatment onset to convert to having negative sputum smears after 2 months of intensive therapy.

OTHER OUTCOMES:
Number of participants lost to follow up during therapy | 6 months
  Lost to follow up is defined as discontinuing treatment for two or more consecutive months (8 weeks) for non-medical reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Pranay Sinha, MD, Principal Investigator — Boston Medical Center; Kobto G Khoura, MD, PhD, Study Director — The International Union Against Tuberculosis and Lung Disease
Locations (2):
- Centre Hospitalier et Universitaire de Pneumo-phtisiologie, Porto-Novo, Benin
- National Tuberculosis Programme, Lomé, Togo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cintron C, Dauphinais M, Fiogbe AA, Dogo MF, Ate S, Adjonou C, Agossou K, Pan SJ, Esse M, Ade B, Adjoh KS, Affolabi D, Sinha P, Koura KG. Impact of Nutritional Support for Tuberculosis on Intermediate and Terminal Undernutrition and Treatment Outcomes (INSTITUT) study: a protocol for a quasi-experimental study to assess the impact of nutritional support on tuberculosis treatment outcomes in Benin and Togo. BMJ Open. 2025 Feb 10;15(2):e088629. doi: 10.1136/bmjopen-2024-088629. PMID 39929516